CLINICAL TRIAL: NCT06504407
Title: BINGO: Bridging Knowledge, Increasing Awareness - Empowering the Black Community Through Educational Gamification on Cancer Screenings and Clinical Trial Diversity
Brief Title: BINGO: Bridging Knowledge, Increasing Awareness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Monali Vasekar, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PSCI-24-021
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer Education; Health Equity

STUDY DESIGN:
Intervention Model Description: Single arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bingo Educational Intervention (Experimental): Single-arm, interventional study where all participants will engage in the Bingo game as an educational intervention.
  Interventions: Behavioral: Bingo Educational Game

INTERVENTIONS:
Behavioral: Bingo Educational Game — The intervention involves Bingo games designed to educate African American/Black community members about cancer and clinical trials. During each game, educational facts are shared, and prizes promoting healthy lifestyles are awarded. Led by a Diversity Navigator, the sessions include pre- and post-test surveys to assess knowledge gain and engagement. The intervention also connects participants with needed medical services.

SUMMARY:
The U.S. population is becoming more diverse, but minority groups are still significantly underrepresented in cancer clinical trials. This disparity limits our understanding of how treatments work across different populations. Efforts like the 21st Century Cures Act aim to improve inclusion, but challenges persist due to historical mistrust and complex barriers in healthcare.

To address these issues, Penn State Health is using a fun and educational approach called "BINGO" to engage the African American/Black community in Dauphin and surrounding counties. Led by the PSCI Diversity Navigator, these BINGO games will provide information about cancer and clinical trials in a relaxed setting. The goal is to build trust, increase awareness, and ultimately improve participation of underrepresented groups in clinical trials.

Through this initiative, they hope to connect participants with needed healthcare services and gather feedback to tailor future trials to community needs. This approach aims to foster collaboration between minority communities and the healthcare system, ensuring that clinical trials reflect the diversity of the population they aim to serve.

DETAILED DESCRIPTION:
Penn State Health is addressing the underrepresentation of minority groups in cancer clinical trials through a community-engagement initiative using a BINGO educational game. Despite efforts like the 21st Century Cures Act, minority participation remains low, impacting the generalizability of trial results and access to novel treatments for diverse populations.

Led by the PSCI Diversity Navigator, this initiative focuses on the African American/Black community in Dauphin and surrounding counties. The BINGO games serve as a platform to educate participants about cancer, clinical trials, and the importance of diversity in research. By creating a relaxed and enjoyable atmosphere, the initiative aims to build trust and increase awareness among community members.

The project's long-term goals include fostering collaboration between minority communities and Penn State Health, improving clinical trial participation rates among underrepresented populations, and addressing healthcare disparities. Immediate objectives involve assessing the feasibility, educational utility, and engagement of the BINGO game through pre- and post-game surveys and knowledge tests.

Recruitment efforts target community centers and organizations like historically Black sororities and churches, leveraging their influence and trust within the community. The initiative strategically focuses on areas with high African American populations, such as Harrisburg, to maximize impact and engagement.

Feedback gathered from participants will guide future trial designs tailored to community needs, enhancing the inclusivity and relevance of research efforts. By promoting understanding and trust, Penn State Health aims to create a model that can be replicated to improve minority participation in clinical trials nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults aged 18 years and above.
2. Gender Identity: Individuals identifying as cisgender, transgender, or females.
3. Language Proficiency: Proficiency in English equivalent to middle school/high school level.
4. Registration: Completion of registration via the provided RedCap link prior to the Bingo session.
5. Consent: Willingness to provide written consent at the beginning of the Bingo session to participate in the research study.

Exclusion Criteria:

1. Age: Individuals under the age of 18 years.
2. Gender Identity: Participants who do not identify as cisgender, transgender, or females.
3. Language Proficiency: Inability to understand English at a middle school/high school level.
4. Previous Participation: Individuals who have already participated in a previous Bingo game session for this study.
5. Medical or Cognitive Impairment: Participants unable to provide informed consent or actively participate due to medical or cognitive reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-12-13 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measure | one year
  Percentage of Participants Attending a Complete Bingo Game Session and Completing Pre- and Post-Test Surveys.
Utility Measure | one year
  Pre- and post-test scores on knowledge-based questions will be compared to measure the effectiveness of the educational content.
Engagement Measure | one year
  Participant engagement will be evaluated using a 5-point Likert scale, with the percentage of participants who "strongly agree or agree" that Bingo game was engaging being the primary measure.

CONTACTS AND LOCATIONS:
Overall Officials: Monali Vasekar, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Information will be collected in De identified manner . IPD will not be shared with any other researchers.